CLINICAL TRIAL: NCT06195514
Title: Expanded Access Program: Fruquintinib for Patients With Metastatic Colorectal Cancer Who Progressed After Standard Therapy
Brief Title: Expanded Access to TAK-113 for Adults With Metastatic Colorectal Cancer (mCRC)
Status: No longer available | Type: Expanded Access
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-113 EAP
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Drug Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: TAK-113 — Description: TAK-113 5 mg capsules, orally, once daily, in a 3 weeks on/1 week off schedule for each 4-week cycle per treatment guidelines.
  Other Names: Fruquintinib; HMPL-013

SUMMARY:
The expanded access program allows people to gain access to an unlicensed treatment on compassionate grounds. This expanded access program provides adults with refractory metastatic colorectal cancer (mCRC) and who cannot neither adequately be treated by current standard of care nor participate in a clinical study access to TAK-113 until TAK-113 becomes commercially available in the respective country or the adult does no longer seem to benefit from treatment with TAK-113.

DETAILED DESCRIPTION:
This is an expanded access program in which the drug being given is called TAK-113. This study will provide early access to TAK-113 until commercial availability in the respective country, for eligible participants with refractory mCRC who cannot adequately be treated by current standard of care and who cannot enter a clinical trial.

All participants will receive TAK-113 5 mg oral capsules in a 3 weeks on/1 week off schedule for each 4-week cycle.

As a part of the expanded access program, there will be a voluntary non-interventional real-world data collection of information.

This is a multi-center international program. Participants will continue treatment until disease progression, unacceptable toxicity, withdrawal of consent, the treatment becomes commercially available, or halting of product development.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) physical status of 0-2.
2. Histologically and/or cytologically documented metastatic colorectal adenocarcinoma.
3. Received all locally available and appropriate prior standard therapies and no other satisfactory treatment option is available for this condition. Participants may have received either prior TAS-102 or regorafenib. Must have progressed on or intolerant to fluoropyrimidine-, oxaliplatin-, and irinotecan- based chemotherapies, anti-vascular endothelial growth factor (VEGF) therapy, and, if rat sarcoma (RAS) wild-type, an anti- epidermal growth factor receptor (EGFR) therapy if available locally for this condition.
4. Adequate bone marrow and organ function as defined by the following:

   1. Absolute neutrophil count of ≥1.5×10^9 per liter, platelet count of ≥75×10^9 per liter, and hemoglobin ≥8 grams per deciliter (g/dL).
   2. Serum total bilirubin ≤1.5 times the upper limit of normal (ULN)
   3. Urine dipstick ≤1+ for proteinuria or ≤30 milligrams per deciliter (mg/dL) in urinalysis, unless quantitative protein is <1000 milligram (mg) in a 24-hour urine sample or urine protein: creatinine ratio on spot urine testing is ≤1.9.
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase levels ≤2.5 times the ULN (participants with liver metastases must have ALT and AST levels ≤5 times the ULN).
   5. Serum creatinine ≤1.5 times the ULN or creatinine clearance ≥60 milliliters per minute (mL/min).
5. Ineligible for other clinical trials of investigational drugs for refractory mCRC, if available.

Exclusion Criteria:

1. Received systemic anticancer therapies [including chemotherapy, tyrosine-kinase inhibitors (TKIs) and endocrine therapy] within 2 weeks prior to the first dose of study drug.

   NOTE: If participant is currently receiving TAK-113 outside of a clinical trial and benefitting from treatment, they may still be considered provided they meet all other criteria.
2. Uncontrolled hypertension as defined per local institution.
3. Any unresolved toxicities from a previous antitumor treatment greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 grade 1 (except for alopecia or neurotoxicity grade≤2).
4. Major surgery within the last 60 days or have had any other minor surgery or invasive procedure within the last 4 weeks.
5. Any thromboembolic events (including deep vein thrombosis, and pulmonary embolism) within the past 6 months, or history of stroke and/or transient ischemic attack within the last 12 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/674b1cc207334911??page=1&idFilter=TAK-113+EAP